CLINICAL TRIAL: NCT03075852
Title: Comparative Analysis of Three-dimensional Heads-up Display Surgical Platform to Standard Operating Microscope for Vitreoretinal Surgery
Brief Title: Comparision of Retinal Surgery by Three-dimensional Heads-up Display to the Standard Operating Microscope
Status: Completed | Type: Observational
Sponsor: MidAtlantic Retina (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, MidAtlantic Retina, Investigator, Wills Eye
Organization: Wills Eye (Other)
Other Study IDs: 17-609E
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Comparison of 3D Visualization and Microscope for VR Surgery
Keywords: Heads-up display, NGENUITY, Vitreoretinal surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- 3D VRS Patients: Those who undergo surgery with NGENUITY (3D VRS-Vitreoretinal surgery)
  Interventions: Device: Heads- Up Display Surgery
- Standard operating microscope: Those who undergo surgery with the standard operating microscope

INTERVENTIONS:
Device: Heads- Up Display Surgery — Patient undergoes VR surgery with visualization using heads up display 3D monitor viewed by the operating surgeon.
  Other Names: NGENUITY surgical display system
  Groups: 3D VRS Patients

SUMMARY:
Prospective, cross-sectional, observational study investigating a three dimensional heads up display for retinal surgery and comparing its outcomes and ease of use with the standard operative microscope.

DETAILED DESCRIPTION:
Prospective, cross-sectional, observational study. Patient are undergoing vitreoretinal surgery for a variety of indications including, but not limited to, epiretinal membrane (ERM), macular hole, vitreous opacities, vitreous hemorrhage, aphakia, dislocated or displaced intraocular or crystalline lens, rhegmatogenous retinal detachment, and tractional retinal detachment. In this prospective, single-center, unmasked cross-sectional, observational case series, at minimum of 100 consecutive eyes will undergo 23-, 25-, or 27-gauge 3-port pars plana vitrectomy (PPV) with the Constellation Vision System (Alcon Laboratories, Hünenberg, Switzerland) using either the NGENUITY 3D HUD surgery platform or standard operating microscope (OPMI Lumera 700 surgical microscope with ReSight (Carl Zeiss AG, Gena, Germany), with 1:1 randomization. Surgical gauge will be dictated by operating surgeon preference. Informed consent will be obtained from all patients enrolled in accordance with the Declaration of Helsinki and all applicable HIPPA regulations. All surgeries will be digitally recorded (as is routinely done for educational purposes) and video data will be stored on password-protected, encrypted external hard-disk drives. These drives will be stored in a secure, locked cabinet in the Research Department of the Retina Service when not in use. All surgeries will be performed by 2 surgeons (AH and JH). Those randomized to 3D HUD surgery will undergo PPV with a 3D high dynamic range camera (ICM5), specialized image processing software (Version 9.5.4; TrueWare, Santa Barbara, CA), and a 46" high-definition (1980x1024 pixel) liquid crystal display (GD-463D10, Yokohama, Japan). During surgery with the 3D HUD, the surgeon will wear passive 3-D polarized glasses and will be positioned approximately 1.5 m from the display. Iris aperture and image gain will be standardized and unchanged for all cases performed with the 3D HUD. Enrolled patients will be monitored at post-operative day 1, week 1, month 1, and month 3 to measure visual acuity, undergo optical coherence tomography (OCT) if clinically indicated, and further examination to document anterior segment and dilated funduscopic examination findings. Patients undergoing epiretinal membrane (ERM) and internal limiting membrane (ILM) removal for either macular pucker or macular hole repair will be subjected to a disease-specific surgical protocol to examine potential differences in macular surgery between 3D HUD and traditional microscope visualization. These patients will undergo 25-gauge 3-port PPV with 1:1 randomization to either visualization with the 3D HUD or standard operating microscope. Indocyanine green (ICG) vital dye (**% solution) will be injected in 0.1 cc aliquots to stain the ILM with the infusion cannula clamped and 60 seconds allowed for the dye to stain the ILM. Endoillumination levels will initially be set to 1% and will be increased by 1% intervals until the operating surgeon notes enough illumination to proceed with ERM/ILM peeling. ILM peeling will be performed to the boundaries of the retinal vascular arcades and the duration of membrane peeling will be documented. If the operating surgeon requests increased endoilluminaton power during membrane peeling, the increased value will be recorded. The number of macular hemorrhages and contusions induced by direct forcep trauma as well as iatrogenic retinal breaks sustained during membrane peeling will also be recorded. Data Collection Demographic data, diagnosis, clinical presentation, and history will be recorded for each patient on initial examination as is done in the course of routine care. Data elements will include age, race, date of birth, date of evaluation, medical record number, chief complaint, past ocular history, past medical history, visual acuity, anterior segment exam findings (i.e. ocular surface disease, lens status, etc.), funduscopic exams, preoperative imaging and testing (OCT, FAF, Fundus Photography). Intraoperative endoillumination levels will be recorded. Recorded surgical video files and follow-up status will be compiled for each patient and various metrics will be recorded including total operative time, time of ILM/ERM peeling, number of ICG aliquots required to visualize the ILM, and intraoperative complications. Baseline and follow up data will also include visual acuity, anterior segment and funduscopic examination, and OCT data if applicable. Other data collected will include subjective physician surveys on the use of the two visualization systems, including quality of visualization on a 10-point scale, perceived subjective difficulties with vitreoretinal visualization, and overall ergonomic comfort on a 10-point scale. Human Subjects and Informed Consent The tenets of the Declaration of Helsinki will be followed and written informed consent obtained at the time of patient enrollment. Patients will also be provided with a lay explanation of the study goals and protocol. The decision to enroll in the study is entirely elective and patients will not be reimbursed for their participation. The PHI and privacy of subjects will be maintained by strict adherence to HIPPA and Wills Eye Institute policies. The aforementioned data will be stored prospectively as patients are enrolled. All data upon collection will be coded and de-identified. Codes will be created for each consecutive patient via a random number generator. All data will be stored on a computer stored and ecrypted hard drives within an ecrypted password protected Microsoft Excel file only accessible to members of the study team. De-identified data will be linked to medical record numbers and date of birth. No other patient identifiers will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those age 18 or older undergoing vitreoretinal surgery for a variety of indications including, but not limited to, epiretinal membrane (ERM), macular hole, vitreous opacities, vitreous hemorrhage, aphakia, dislocated or displaced intraocular or crystalline lens, rhegmatogenous retinal detachment, and tractional retinal detachment

Exclusion Criteria:

* Prisoners, institutionalized patients, and those who have undergone previous pars plana vitrectomy will be excluded. Patients undergoing combined, simultaneous scleral buckle placement and pars plana vitrectomy will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those age 18 or older undergoing vitreoretinal surgery from the Mid Altantic Retina, Wills Eye location office, for a variety of indications including, but not limited to, epiretinal membrane (ERM), macular hole, vitreous opacities, vitreous hemorrhage, aphakia, dislocated or displaced intraocular or crystalline lens, rhegmatogenous retinal detachment, and tractional retinal detachment
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Intraoperative complications | day of surgery
  Intraoperative complications including: increased surgical time, needing to switch to standard operating microscope, increased time for ILM/ ELM peeling

SECONDARY OUTCOMES:
Visual Acuity | baseline and 3 months
  Snellen

OTHER OUTCOMES:
Intraoperative time | day of surgery
  Duration of surgery
Ease of use score | day of surgery
  Physician ease-of-use score on a 10 point scale to quantify usability of 3D HUD and standard operating scope.

CONTACTS AND LOCATIONS:
Overall Officials: Allen C Ho, MD, Principal Investigator — Mid Atlantic Retina
Locations (1):
- MidAtlantic Retina-Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckardt C, Paulo EB. HEADS-UP SURGERY FOR VITREORETINAL PROCEDURES: An Experimental and Clinical Study. Retina. 2016 Jan;36(1):137-47. doi: 10.1097/IAE.0000000000000689. PMID 26200516